CLINICAL TRIAL: NCT01100112
Title: Multicenter, Open-Label Efficacy and Safety Study of Oral Budesonide-MMX 9mg Extended Release Tablets in Patients With Mild to Moderate, Active Ulcerative Colitis
Brief Title: (CB-01-02/06) Oral Budesonide-Multi-Matrix System (MMX) 9mg Extended Release Tablets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-01-02/06
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Colitis, Ulcerative
Keywords: ulcerative colitis; Budesonide
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Budesonide (Experimental): Budesonide-MMX 9 mg tablet
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — One Budesonide-MMX 9 mg tablet will be taken in the morning after breakfast for 8 weeks.

SUMMARY:
Open-label, 8 week study, to assess the efficacy and safety of oral Budesonide-MMX 9 mg Extended-release Tablets in patients with mild to moderate, active ulcerative colitis who are not in remission based on the Ulcerative Colitis Disease Activity Index in study CB-01-02/01 (parent study [NCT00679432]).

DETAILED DESCRIPTION:
Patients who complete the parent study and who do not achieve clinical remission will be eligible to receive 8 weeks of open-label treatment with Budesonide-MMX 9mg if they satisfy the entry criteria for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 74 years of age, who are able to understand and voluntarily provide written informed consent
* Completed all Final Visit assessments for study CB-01-02/01 (NCT00679432) and are not in clinical remission
* Diagnosis of ulcerative colitis of mild to moderate severity with an Ulcerative Colitis Disease Activity Index (UCDAI) <or= 10 according to Sutherland
* Females of child-bearing potential must have had a serum pregnancy test performed at the Final Visit of the parent study, and must use an acceptable contraceptive method throughout the treatment period. Female subjects must also not be actively breast-feeding through the entire study period.
* Ability to comprehend the full nature and purpose of the study, including possible risks and side effects
* Ability to co-operate with the investigator and to comply with the requirements of the entire study

Exclusion Criteria:

* Did not complete study CB-01-02/01
* Achieved clinical remission in study CB-01-02/01
* Patients with severe ulcerative colitis (UCDAI >10)
* Patients with infectious colitis
* Evidence or history of toxic megacolon
* Severe anemia, leucopenia, or granulocytopenia
* Use of immunosuppressive agents in the last 8 weeks before the study
* use of anti-tumor necrosis factor alpha agents in the last three months
* Concomitant use of any rectal preparation for the treatment of ulcerative colitis
* Concomitant use of antibiotics
* Concurrent use of cytochrome P-450 3A4 (CYP3A4) inducers and CYP3A4 inhibitors.
* Patients with verified, presumed of expected pregnancy or ongoing lactation
* Patients with liver cirrhosis, or evident hepatic or renal disease or insufficiency and/or severe impairment of the bio-humoral parameters (i.e., 2x upper limit of normal for alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transpeptidase, or creatinine)
* Patients with severe disease(s) in other organs of systems
* Patients with local of systemic complications of other pathological states requiring a therapy with corticosteroids and/or immunosuppressive agents
* Patients diagnosed with Type 1 diabetes
* Patients diagnosed with or with a family history of glaucoma
* Patients with known hepatitis B, hepatitis C, or with human immunodeficiency virus (HIV), according to the local privacy policy
* Any other medical condition that in the principal investigator's opinion would make the administration of the study drug or study procedures hazardous to the subject or obscure the interpretation of adverse events

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- India (15):
  - Santarus Clinical Investigational Site 9001, Andhra Pradesh
  - Santarus Clinical Investigational Site 9009, Andhra Pradesh
  - Santarus Clinical Investigational Site 9012, Andhra Pradesh
  - Santarus Clinical Investigational Site 9016, Andhra Pradesh
  - Santarus Clinical Investigational Site 9006, Assam
  - Santarus Clinical Investigational Site 9007, Gujarat
  - Santarus Clinical Investigational Site 9004, Karnataka
  - Santarus Clinical Investigational Site 9015, Karnataka
  - Santarus Clinical Investigational Site 9003, Kerala
  - Santarus Clinical Investigational Site 9002, Maharashtra
  - Santarus Clinical Investigational Site 9008, Maharashtra
  - Santarus Clinical Investigational Site 9013, Maharashtra
  - Santarus Clinical Investigational Site 9018, Rajasthan
  - Santarus Clinical Investigational Site 9005, Tamil Nadu
  - Santarus Clinical Investigational Site 9014, Uttar Pradesh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from February 2010 to July 2010
Pre-assignment Details: Patient had to have failed to achieve clinical remission in parent study CB-01-02/01. One of the 61 enrolled patients did not receive study drug. Therefore, 60 patients were evaluable for safety and efficacy analyses.
Groups:
- Budesonide: Budesonide-multi-matrix system (MMX) 9 mg tablet
  Budesonide : One Budesonide-MMX 9 mg tablet will be taken in the morning after breakfast for 8 weeks.
Period: Overall Study
Arm/Group | Budesonide
Started | 60
Completed | 52
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: All patients who received at least 1 dose of study drug were considered Evaluable patients. Total evaluable population was 60.
Groups:
- Budesonide: Budesonide-MMX 9 mg tablet
  Budesonide : One Budesonide-MMX 9 mg tablet will be taken in the morning after breakfast for 8 weeks.
Arm/Group | Budesonide
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Region of Enrollment [Number; unit: participants]
  India | 60

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Achieving Clinical Remission
Description: The primary efficacy endpoint is clinical remission at 8 weeks, defined as a Ulcerative Colitis Disease Activity Index score of < or = 1 with a score of 0 for both rectal bleeding and stool frequency, and > or = 1 point reduction from baseline in endoscopy score, without any sign of mucosal friability (a score of 0 for mucosal appearance).
  The UCDAI has 4 components. Each component is scored on scale of 0 to 3 (total maximum [worst] score = 12). Definitions of component scores are as follows: stool frequency: 0 = normal frequency, 1 = 1 - 2 stools per day greater than normal frequency, 2 = 3 - 4 stools per day greater than normal frequency, and 3 = > 4 stools per day greater than normal frequency; rectal bleeding: 0 = none, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood; physician's rating of disease activity: 0 = normal, 1 = mild, 2 = moderate, 3 = severe; mucosal appearance: 0 = normal, 1 = mild friability, 2 = moderate friability, 3 = exudation, spontaneous bleeding.
Time Frame: At the end of the 8 week treatment period
Population: All patients who received at least 1 dose of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Budesonide
Number analyzed (Participants) | 60
percentage of patients | 25

2. Secondary Outcome: The Secondary Efficacy Endpoint is Clinical Improvement
Description: The secondary efficacy endpoint is clinical improvement, defined as a drop in the Ulcerative Colitis Disease Activity Index score of > or = 3 points from baseline.
Time Frame: After 8 weeks treatment period
Population: All patients who received at least 1 dose of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Budesonide
Number analyzed (Participants) | 60
percentage of patients | 26.7

3. Secondary Outcome: Safety Evaluations: the Numbers of Patients Who Experience Serious Adverse Events (SAEs) or Other Nonserious Adverse Events (AEs) During the Course of the Study.
Description: Safety will be assessed by evaluating SAEs and AEs. The outcome measure data are the numbers of patients who experienced SAEs or other nonserious AEs.
Time Frame: Throughout the 8 week treatment period
Population: All patients who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Budesonide
Number analyzed (Participants) | 60
participants
  Serious Adverse Events | 2
  Other non-serious adverse events | 29

4. Secondary Outcome: Endoscopic Improvement
Description: Greater or equal to a 1 point improvement in the mucosal appearance subscore of the ulcerative colitis disease activity index (UCDAI), from baseline to week 8.
  The UCDAI mucosal appearance subscore is graded as follows: 0 = normal, 1 = mild friability, 2 = moderate friability, 3 = exudation, spontaneous bleeding.
Time Frame: 8 weeks
Population: All patients who received at least one dose of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Budesonide
Number analyzed (Participants) | 60
percentage of patients | 40

ADVERSE EVENTS:
Time Frame: 56 day ± 2 day (study duration) + 30 day safety followup period.
Arm/Group | Budesonide
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 29/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide (N=60)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide (N=60)
Cushingoid (Endocrine disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7)
Blood cortisol decreased (Investigations) | 9 (9)
Blood glucose decreased (Investigations) | 2 (2)
Blood potassium increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
This was an open label study. There was no reference therapy for statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No